CLINICAL TRIAL: NCT01660477
Title: A Phase 1, Open-Label, Parallel Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of Multiple Doses of Lopinavir/Ritonavir and the Effects of Lopinavir/Ritonavir on the Pharmacokinetics of Multiple Doses of Isavuconazole in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study Between Lopinavir/Ritonavir and Isavuconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 9766-CL-0035
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Lopinavir/Ritonavir; Healthy Volunteers
Keywords: Isavuconazole; Lopinavir/ritonavir; Healthy Volunteers; BAL8557; Kaletra ®
MeSH Terms: interventions — isavuconazole; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: isavuconazole only (Experimental): Isavuconazole three times per day (TID) on Days 1-2, and once daily (QD) on Days 3 thru 13
  Interventions: Drug: Isavuconazole
- Arm 2 : LPV/RTV only (Experimental): Lopinavir/ritonavir (LPV/RTV) twice daily (BID) on Days 1-12 and once on Day 13
  Interventions: Drug: Lopinavir/ritonavir
- Arm 3: isavuconazole and LPV/RTV (Experimental): Isavuconazole three times per day (TID) on Days 1-2, and once daily (QD) on Days 3 thru 13 in combination with lopinavir/ritonavir twice daily (BID) on Days 1-13
  Interventions: Drug: Isavuconazole; Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL8557
  Arms: Arm 1: isavuconazole only; Arm 3: isavuconazole and LPV/RTV
Drug: Lopinavir/ritonavir — oral
  Other Names: KALETRA®
  Arms: Arm 2 : LPV/RTV only; Arm 3: isavuconazole and LPV/RTV

SUMMARY:
The purpose of this two part study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of multiple doses of lopinavir/ritonavir and the effect of multiple doses of lopinavir/ritonavir on the pharmacokinetics of isavuconazole.

Part 1 of the study includes 12 subjects randomized to receive either isavuconazole alone or isavuconazole in combination with lopinavir/ritonavir. The purpose of Part 1 is to evaluate safety and tolerability and to establish the effect of multiple doses of lopinavir/ritonavir on isavuconazole.

Part 2, if initiated, includes 54 subjects randomized to receive isavuconazole alone, lopinavir/ritonavir alone, or isavuconazole in combination with lopinavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT), total bilirubin, lipase, amylase, glucose and triglycerides must be within the normal range
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a history of pancreatitis
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including lopinavir/ritonavir or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions- - The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen
* The subject has participated in a previous isavuconazole study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) for isavuconazole: AUCtau | Part 1, Day 13: predose, 0.5, 1, 2, 3, 4, 6, 8,10,12,16, and 24 hours post-dose
  (Arms 1 and 3) Area under the concentration time curve during the during time interval between consecutive dosing (AUCtau) (tau=24)
Pharmacokinetic (PK) profile for isavuconazole: AUC tau and Cmax | Part 2, Day 13: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours post dose
  (Arms 2 and 3) Maximum concentration (Cmax)
Pharmacokinetic (PK) profile for lopinavir/ritonavir: AUC tau and Cmax | Part 2, Day 13: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours post dose
  (Arms 2 and 3) AUC during time interval between consecutive dosing (AUCtau) (tau=12)

SECONDARY OUTCOMES:
PK for isavuconazole (in plasma): trough concentration (Ctrough) | Parts 1 and 2, Days 3, 5, 7, 9 and 11: pre-dose
  (Arms 1 and 3)
PK profile for isavuconazole (in plasma): Cmax, tmax | Parts 1 and 2, Day 13: predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12,16, and 24 hours post-dose
  (Arms 1 and 3) Time to attain Cmax (tmax)
PK for lopinavir/ritonavir (in plasma): trough concentration (Ctrough) | Part 2, Days 3, 5, 7, 9 and 11: pre-dose
  (Arms 2 and 3)
PK for lopinavir/ritonavir (in plasma): tmax | Part 2, Day 13: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours post dose
  (Arms 2 and 3)
Safety and tolerability of isavuconazole alone and in combination with lopinavir (LPV) and ritonavir (RTV) assessed by recording of adverse events, physical examination, clinical laboratory evaluation, electrocardiograms (ECGs) and vital signs | Part 1, Days 1 - 20 ± 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, Glendale, California, United States